CLINICAL TRIAL: NCT04414995
Title: Effect of Paracetamol and Ibuprofen When Intravenously Given Combination or Alone in Reducing Morphine Requirements After Total Knee Arthroplasty
Brief Title: Effect of Paracetamol and Ibuprofen Reducing Morphine Requirements After Total Knee Arthroplasty
Acronym: PctIbfFKUI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andri Maruli Tua Lubis, Head of Research Division RSCM, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Pct-Ibf-FKUI
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Analgesia
Keywords: multi modal analgesia
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Ibuprofen; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients in Group 1 received a combination of 1000 mg IV paracetamol and 800 mg IV ibuprofen at the end of operation followed by 1000 mg IV paracetamol and 800 mg IV ibuprofen every 6 hours up to 72 hours.
  Patients in Group 2 received 1000 mg IV paracetamol and 100 ml IV normal salines at the end of operation followed by 1000 mg IV paracetamol and 100 ml IV normal salines every 6 hours up to 72 hours.
  Patients in Group 3 received 800 mg IV ibuprofen and 100 ml IV normal salines at the end of operation followed by 800 mg IV ibuprofen and 100 ml IV normal salines every 6 hours up to 72 hours.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study medication will be masked by the pharmacy. Participants, those administrating the intervention, other caregivers, outcome assessors, data managers, statisticians, and investigators drawing conclusions will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Paracetamol+Ibuprofen (Experimental): Patients in Group 1 will receive a combination of 1000 mg IV paracetamol and 800 mg IV ibuprofen at the end of operation following by 1000 mg IV paracetamol and 800 mg IV ibuprofen every 6 hours up to 72 hours.
  Interventions: Drug: Paracetamol injection and Ibuprofen injection
- Paracetamol+normal saline (Experimental): Patients in Group 2 will receive 1000 mg IV paracetamol and 100 ml IV normal salines at the end of operation following by 1000 mg IV paracetamol and 100 ml IV normal salines every 6 hours up to 72 hours.
  Interventions: Drug: Paracetamol injection and normal saline
- Ibuprofen+normal saline (Experimental): Patients in Group 3 will receive 800 mg IV ibuprofen and 100 ml IV normal salines at the end of operation following by 800 mg IV ibuprofen and 100 ml IV normal salines every 6 hours up to 72 hours.
  Interventions: Drug: Ibuprofen Injection and normal saline

INTERVENTIONS:
Drug: Paracetamol injection and Ibuprofen injection — Use of combination acetaminophen and ibuprofen to reduce morphine requirement inpatient after Total knee arthroplasty
  Other Names: Paracetamol and Ibuprofen
  Arms: Paracetamol+Ibuprofen
Drug: Paracetamol injection and normal saline — Use of paracetamol and normal saline to reduce morphine requirement inpatient after Total knee arthroplasty
  Other Names: Paracetamol injection
  Arms: Paracetamol+normal saline
Drug: Ibuprofen Injection and normal saline — Use of ibuprofen and normal saline to reduce morphine requirement inpatient after Total knee arthroplasty
  Other Names: Ibuprofen injection
  Arms: Ibuprofen+normal saline

SUMMARY:
Adequate pain management has an important role in supporting early ambulation after the Total Knee Arthroplasty (TKA). Multimodal analgesia is one of the modalities of overcoming postoperative pain. The use of combination Paracetamol and Ibuprofen injection is expected to reduce total morphine consumption after TKA.

DETAILED DESCRIPTION:
The research will compare the effect of paracetamol injection and ibuprofen injection when given alone or in combination to reduce morphine requirement in a patient after total knee arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with 20 < BMI < 30 kg/m2
* Adult patient with knee varus alignment 10-20°

Exclusion Criteria:

* Impaired cardiac, liver, and/or renal function.
* History of substance abuse or chronic pain.
* Patients are known to be hypersensitive to any of the components of IV ibuprofen or IV paracetamol.
* Patients currently on anticoagulation medications.
* Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board) and agree to abide by the study restrictions.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Total morphine requirement | 24 hours
  morphine requirement in patient after total knee arthroplasty procedure

SECONDARY OUTCOMES:
Numerical rating scale of pain in resting phase, walking phase, knee full flexion phase | 24 hours, 48 hours, 72 hours
  amount of pain measure by numerical rating scale. Patients rate their pain from 0 to 10, Zero represents "no pain," whereas 10 represents the opposite end of the pain continuum (e.g., "the most intense pain imaginable," "pain as intense as it could be," "maximum pain")
range of motion knee in flexion and extension | 24 hours, 48 hours, 72 hours
  range of motion knee in flexion and extension
2MWT after total knee arthroplasty procedure | 24 hours, 48 hours, 72 hours
  amount of walking length in 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Andri MT Lubis, MD, PhD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia; Aida R Tantri, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia; Ludwig AP Pontoh, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (2):
- Indonesia (2):
  - Fatmawati General Hospital, Jakarta, DKI Jakarta
  - Cipto Mangunkusumo National General Hospital, Jakarta Pusat, DKI Jakarta

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan (SAP)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: data will become available after study completion.
Access Criteria: others researches contact

REFERENCES:
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Affas F, Nygards EB, Stiller CO, Wretenberg P, Olofsson C. Pain control after total knee arthroplasty: a randomized trial comparing local infiltration anesthesia and continuous femoral block. Acta Orthop. 2011 Aug;82(4):441-7. doi: 10.3109/17453674.2011.581264. Epub 2011 May 11. PMID 21561303
- [Background] Barrington JW, Lovald ST, Ong KL, Watson HN, Emerson RH Jr. Postoperative Pain After Primary Total Knee Arthroplasty: Comparison of Local Injection Analgesic Cocktails and the Role of Demographic and Surgical Factors. J Arthroplasty. 2016 Sep;31(9 Suppl):288-92. doi: 10.1016/j.arth.2016.05.002. Epub 2016 May 12. PMID 27318410
- [Background] Oderda GM, Gan TJ, Johnson BH, Robinson SB. Effect of opioid-related adverse events on outcomes in selected surgical patients. J Pain Palliat Care Pharmacother. 2013 Mar;27(1):62-70. doi: 10.3109/15360288.2012.751956. Epub 2013 Jan 9. PMID 23302094
- [Background] Sharma V, Morgan PM, Cheng EY. Factors influencing early rehabilitation after THA: a systematic review. Clin Orthop Relat Res. 2009 Jun;467(6):1400-11. doi: 10.1007/s11999-009-0750-9. Epub 2009 Mar 10. PMID 19277807
- [Background] Woolf CJ, Salter MW. Neuronal plasticity: increasing the gain in pain. Science. 2000 Jun 9;288(5472):1765-9. doi: 10.1126/science.288.5472.1765. PMID 10846153
- [Background] Horlocker TT, Kopp SL, Pagnano MW, Hebl JR. Analgesia for total hip and knee arthroplasty: a multimodal pathway featuring peripheral nerve block. J Am Acad Orthop Surg. 2006 Mar;14(3):126-35. doi: 10.5435/00124635-200603000-00003. PMID 16520363
- [Background] Halawi MJ, Grant SA, Bolognesi MP. Multimodal Analgesia for Total Joint Arthroplasty. Orthopedics. 2015 Jul 1;38(7):e616-25. doi: 10.3928/01477447-20150701-61. PMID 26186325
- [Background] Oderda G. Challenges in the management of acute postsurgical pain. Pharmacotherapy. 2012 Sep;32(9 Suppl):6S-11S. doi: 10.1002/j.1875-9114.2012.01177.x. PMID 22956493
- [Background] Barletta JF. Clinical and economic burden of opioid use for postsurgical pain: focus on ventilatory impairment and ileus. Pharmacotherapy. 2012 Sep;32(9 Suppl):12S-8S. doi: 10.1002/j.1875-9114.2012.01178.x. PMID 22956490
- [Background] Buvanendran A. Multimodal Analgesia for Perioperative Pain Management: ASA Refresh Courses Anesthesiol. 2012;40(1):1-6.
- [Background] Rosero EB, Joshi GP. Preemptive, preventive, multimodal analgesia: what do they really mean? Plast Reconstr Surg. 2014 Oct;134(4 Suppl 2):85S-93S. doi: 10.1097/PRS.0000000000000671. PMID 25255012
- [Background] Derry CJ, Derry S, Moore RA. Single dose oral ibuprofen plus paracetamol (acetaminophen) for acute postoperative pain. Cochrane Database Syst Rev. 2013 Jun 24;2013(6):CD010210. doi: 10.1002/14651858.CD010210.pub2. PMID 23794268
- [Background] Dahl JB, Nielsen RV, Wetterslev J, Nikolajsen L, Hamunen K, Kontinen VK, Hansen MS, Kjer JJ, Mathiesen O; Scandinavian Postoperative Pain Alliance (ScaPAlli). Post-operative analgesic effects of paracetamol, NSAIDs, glucocorticoids, gabapentinoids and their combinations: a topical review. Acta Anaesthesiol Scand. 2014 Nov;58(10):1165-81. doi: 10.1111/aas.12382. Epub 2014 Aug 14. PMID 25124340
- [Background] Ong CK, Seymour RA, Lirk P, Merry AF. Combining paracetamol (acetaminophen) with nonsteroidal antiinflammatory drugs: a qualitative systematic review of analgesic efficacy for acute postoperative pain. Anesth Analg. 2010 Apr 1;110(4):1170-9. doi: 10.1213/ANE.0b013e3181cf9281. Epub 2010 Feb 8. PMID 20142348
- [Background] Thybo KH, Hagi-Pedersen D, Wetterslev J, Dahl JB, Schroder HM, Bulow HH, Bjorck JG, Mathiesen O. PANSAID - PAracetamol and NSAID in combination: study protocol for a randomised trial. Trials. 2017 Jan 10;18(1):11. doi: 10.1186/s13063-016-1749-7. PMID 28069072
- [Result] McCartney CJ, Nelligan K. Postoperative pain management after total knee arthroplasty in elderly patients: treatment options. Drugs Aging. 2014 Feb;31(2):83-91. doi: 10.1007/s40266-013-0148-y. PMID 24399578